Version 3 – 05/09/2017 IRAS number: 227681





## An Open Trial of Group Metacognitive Therapy for Anxiety and Depression in Cancer Survivors

## **PARTICIPANT CONSENT FORM**

| Participant Number: | | REC ref: | | | |
|---|---|---|---|---|---|
| | | | | Please li | nitial Box |
| CONSE | ENT FOR PARTIC | CIPATION IN STU | IDY | | |
| I confirm that I have read a above study. I have had the answered satisfactorily. | | | | | |
| I understand that my parti giving any reason, and wit | | | | any time, without | |
| I understand that relevant looked at by regulatory bo Liverpool and Broadgreen permission for these individually be kept confidential, at secure University of Liverpool | dies and/or indivi<br>NHS Trust wher<br>duals to have acc<br>nd that data will o | duals from the Uni<br>e it is relevant to r<br>ess to my records.<br>nly be available th | versity of Liverpool of my taking part in this I understand that my rough restricted, sha | or from the Royal<br>is research. I give<br>by personal details<br>ared areas on the | |
| In the event that I withdraw point of withdrawal to be k | | | for the information o | btained up to the | |
| I agree to take part in the | above-named stu | dy. | | | |
| | ADDITI | ONAL CONSENT | e | | |
| I would like to be informed study in any way. | | | | articipation in the | |
| I agree for the sessions to | be audio recorde | ed | | | |
| I agree that my GP can be informed that I am participating in the above named study | | | | | |
| SIGNATURES Name of Participant | Date | Signa | ture | - | |
| Researcher | Date | <br>Signat | ure | - | |
| Name of person taking consent (If different from researcher) | Date | Signa | ture | - | |